CLINICAL TRIAL: NCT00003830
Title: A Randomized, Phase III Clinical Trial to Compare Sentinel Node Resection to Conventional Axillary Dissection in Clinically Node-Negative Breast Cancer Patients
Brief Title: Surgery to Remove Sentinel Lymph Nodes With or Without Removing Lymph Nodes in the Armpit in Treating Women With Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NSABP Foundation Inc (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSABP B-32; U10CA012027 (NIH); CDR0000066987
Record Dates: First submitted 1999-11-01; First posted 2003-01-28 (Estimated); Results first posted 2017-12-13 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-11

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I: Conventional axillary dissection (Active Comparator): Sentinel node resection immediately followed by axillary dissection
  Interventions: Procedure: conventional surgery
- Arm II: Sentinel node resection followed by node examination (Experimental): Sentinel node resection followed by node examination then axillary dissection if positive sentinel node.
  Interventions: Procedure: Sentinel node resection followed by node examination

INTERVENTIONS:
Procedure: conventional surgery — Sentinel node resection immediately followed by axillary dissection.
  Arms: Arm I: Conventional axillary dissection
Procedure: Sentinel node resection followed by node examination — Sentinel node resection followed by node examination then axillary dissection if positive sentinel node. No axillary dissection for negative sentinel node.
  Arms: Arm II: Sentinel node resection followed by node examination

SUMMARY:
RATIONALE: Removing the sentinel lymph nodes and examining them under a microscope may help plan more effective surgery for breast cancer. It is not yet known if surgery to remove the sentinel lymph nodes is more effective with or without removal of the lymph nodes in the armpit in treating breast cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of surgery to remove the sentinel lymph nodes with or without removal of lymph nodes in the armpit in treating women who have breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the long term control of regional disease by sentinel node resection vs sentinel node resection followed by conventional axillary dissection in women with breast cancer who are clinically node negative and pathologically sentinel node negative.
* Compare the effect of these two regimens on the overall and disease-free survival of these patients.
* Compare the morbidity associated with these two regimens in these patients.
* Compare the prognostic value of these two regimens in patients who are sentinel node negative or positive by pathology.
* Determine whether a more detailed pathology investigation can identify a group of patients with a potentially increased risk of systemic recurrence who are node negative by pathology.
* Determine the technical success rate of sentinel node dissection and the variability of technical success rate in a broad population of surgeons.
* Determine the sensitivity of the sentinel node to determine the presence of nodal metastases in these patients.

Objectives of quality of life questionnaire in sentinel node-negative patients:

* Compare the severity of self-assessed symptoms and activity limitations of patients treated with these two regimens.
* Compare the severity of self-assessed symptoms and activity limitations after breast cancer surgery in patients whose surgery was on the dominant side vs patients whose surgery was on the non-dominant side.
* Compare the impact of arm edema, range of motion, and sensory neuropathy on self-assessed measures of daily functioning, symptoms, and overall quality of life of patients treated with these regimens.

OUTLINE: This is a randomized study. Patients are stratified according to the surgical treatment plan (lumpectomy vs mastectomy), age (49 and under vs 50 and over), and clinical tumor size (no greater than 2.0 cm vs 2.1-4.0 cm vs at least 4.1 cm). Patients are randomized to one of two surgery arms.

All patients receive technetium (Tc 99m) sulfur colloid injected into normal breast tissue within 1 cm of the primary tumor or biopsy cavity and an intradermal injection of technetium (Tc 99m) sulfur colloid, approximately 0.5-8 hours before surgery. Patients also receive an injection of isosulfan blue dye around the tumor or biopsy cavity after a hot spot is identified with a gamma detector. If a hot spot is not identified, the blue dye is injected after a saline bolus injection.

* Arm I: Patients undergo sentinel node resection immediately followed by conventional axillary dissection.
* Arm II: Patients undergo sentinel node resection and an intraoperative examination of sentinel nodes.

Patients with positive sentinel nodes undergo axillary dissection after sentinel node resection.

Patients with cytologically negative sentinel nodes do not undergo axillary dissection.

Patients with cytologically negative but histologically positive sentinel nodes return to surgery for axillary dissection.

Patients with histologically positive sentinel nodes and those in whom the sentinel node is not identified undergo axillary dissection after sentinel node resection.

Patients with pathologically positive, nonaxillary sentinel nodes undergo axillary dissection after sentinel node resection.

Patients with evidence of tumor remaining after surgery undergo a total mastectomy.

Quality of life is assessed at baseline, at weeks 1-3, and then every 6 months for 3 years or until recurrence.

Patients are followed at 1 and 3 weeks, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: Approximately 5,400 patients will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Resectable invasive adenocarcinoma of the breast, confirmed by 1 of the following:

  * Histologically confirmed by core or open biopsy
  * Confirmed by fine needle aspiration cytology AND positive clinical breast examination and ultrasound or mammography
* Clinically negative lymph nodes

  * No positive ipsilateral axillary lymph nodes
  * No prior removal of ipsilateral axillary lymph nodes
  * No suspicious palpable nodes in the contralateral axilla or palpable supraclavicular or infraclavicular nodes, unless proven nonmalignant by biopsy
* No ulceration, erythema, infiltration of the skin or underlying chest wall (complete fixation), peau d'orange, or skin edema of any magnitude

  * Tethering or dimpling of the skin or nipple inversion allowed
* No bilateral malignancy or mass in the opposite breast that is suspicious for malignancy, unless proven nonmalignant by biopsy
* No diffuse tumors or multiple malignant tumors in different quadrants of the breast
* No other prior breast malignancy except lobular carcinoma in situ
* No prior or concurrent breast implants
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 years and older

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* Not specified

Life expectancy:

* At least 10 years (excluding diagnosis of cancer)

Hematopoietic:

* Not specified

Hepatic:

* No hepatic systemic disease

Renal:

* No renal systemic disease

Cardiovascular:

* No cardiovascular systemic disease

Other:

* No prior malignancy within past 5 years except:

  * Effectively treated squamous cell or basal cell skin cancer
  * Surgically treated carcinoma in situ of the cervix
  * Surgically treated lobular carcinoma in situ of the ipsilateral or contralateral breast
* No concurrent psychiatric or addictive disorder

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior immunotherapy for this cancer

Chemotherapy:

* No prior chemotherapy for this cancer, including neoadjuvant chemotherapy

Endocrine therapy:

* No prior hormonal therapy for this cancer

Radiotherapy:

* No prior radiotherapy for this cancer

Surgery:

* See Disease Characteristics
* No prior breast reduction surgery
* Prior excisional biopsy or lumpectomy allowed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5611 (Actual)
Dates: Start 1999-05; Primary Completion 2010-09 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norman Wolmark, MD, Principal Investigator — NSABP Foundation Inc
Locations (78):
- United States (68):
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Sutter Breast Cancer Group, Sacramento, California
  - Kaiser Permanente Medical Center/Kaiser Foundation Hospital - San Diego, San Diego, California
  - Stanford Cancer Center at Stanford University Medical Center, Stanford, California
  - Hartford Hospital, Hartford, Connecticut
  - MBCCOP - Howard University Cancer Center, Washington D.C., District of Columbia
  - Halifax Medical Center, Daytona Beach, Florida
  - Baptist Regional Cancer Institute - Jacksonville, Jacksonville, Florida
  - University of Miami Sylvester Cancer Center, Miami, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - MBCCOP-Cook County Hospital, Chicago, Illinois
  - Creticos Cancer Center at Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Methodist Cancer Center at Methodist Hospital, Indianapolis, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - Stanley S. Scott Cancer Center at Louisiana State University Medical Center - New Orleans, New Orleans, Louisiana
  - Tulane University Medical Center, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Franklin Square Hospital Center, Baltimore, Maryland
  - Cancer Research Center at Boston Medical Center, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center - University Campus, Worcester, Massachusetts
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - CCOP - Beaumont, Royal Oaks, Michigan
  - Providence Cancer Institute at Providence Hospital, Southfield, Michigan
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Methodist Hospital Cancer Center at Nebraska Methodist Hospital - Omaha, Omaha, Nebraska
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - New York Oncology Hematology, P.C. - Albany Regional Cancer Center, Albany, New York
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Akron City Hospital, Akron, Ohio
  - Aultman Hospital Cancer Center at Aultman Health Foundation, Canton, Ohio
  - Jewish Hospital of Cincinnati, Incorporated, Cincinnati, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Reading Hospital and Medical Center, Reading, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Vermont Cancer Center at University of Vermont, Burlington, Vermont
  - Virginia Oncology Associates - Newport News, Newport News, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia
  - Puget Sound Oncology Consortium, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington
  - Camcare Health, Charleston, West Virginia
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
- Canada (9):
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - St. Michael's Hospital - Toronto, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - Royal Victoria Hospital - Montreal, Montreal, Quebec
  - Jewish General Hospital - Montreal, Montreal, Quebec
  - St. Mary's Hospital Center, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec, Quebec
- MBCCOP - San Juan, San Juan, Puerto Rico

REFERENCES:
- [Background] Land SR, Ritter MW, Costantino JP, Julian TB, Cronin WM, Haile SR, Wolmark N, Ganz PA. Compliance with patient-reported outcomes in multicenter clinical trials: methodologic and practical approaches. J Clin Oncol. 2007 Nov 10;25(32):5113-20. doi: 10.1200/JCO.2007.12.1749. PMID 17991930
- [Result] Weaver DL, Le UP, Dupuis SL, Weaver KA, Harlow SP, Ashikaga T, Krag DN. Metastasis detection in sentinel lymph nodes: comparison of a limited widely spaced (NSABP protocol B-32) and a comprehensive narrowly spaced paraffin block sectioning strategy. Am J Surg Pathol. 2009 Nov;33(11):1583-9. doi: 10.1097/PAS.0b013e3181b274e7. PMID 19730364
- [Result] Land SR, Kopec JA, Lee M, et al.: Quality of life in breast cancer patients receiving sentinel-node (SN) biopsy alone or with axillary dissection (AD): results from NSABP protocol B-32. [Abstract] J Clin Oncol 26 (Suppl 15): A-9533, 2008.
- [Result] Julian TB, Anderson SJ, Fourchotte V, et al.: Is completion axillary dissection always required after a positive sentinel node biopsy? NSABP B-32. [Abstract] Breast Cancer Res Treat 106 (1): A-51, S15, 2007.
- [Result] Julian TB, Anderson SJ, Fourchotte V, et al.: Is intraoperative cytology of sentinel nodes useful and predictive for non-sentinel axillary nodes? NSABP B-32. [Abstract] Breast Cancer Res Treat 106 (1): A-3001, 2007.
- [Result] Krag DN, Anderson SJ, Julian TB, Brown AM, Harlow SP, Ashikaga T, Weaver DL, Miller BJ, Jalovec LM, Frazier TG, Noyes RD, Robidoux A, Scarth HM, Mammolito DM, McCready DR, Mamounas EP, Costantino JP, Wolmark N; National Surgical Adjuvant Breast and Bowel Project. Technical outcomes of sentinel-lymph-node resection and conventional axillary-lymph-node dissection in patients with clinically node-negative breast cancer: results from the NSABP B-32 randomised phase III trial. Lancet Oncol. 2007 Oct;8(10):881-8. doi: 10.1016/S1470-2045(07)70278-4. PMID 17851130
- [Result] Julian B, Fourchotte V, Anderson S, et al.: Predictive factors that identify patients not requiring a sentinel node biopsy: continued analysis of the NSABP B-32 sentinel node trial. [Abstract] Breast Cancer Res Treat 100 (Suppl 1): A-2003, S80-1, 2006.
- [Result] Weaver DL, Krag DN, Manna EA, Ashikaga T, Waters BL, Harlow SP, Bauer KD, Julian TB. Detection of occult sentinel lymph node micrometastases by immunohistochemistry in breast cancer. An NSABP protocol B-32 quality assurance study. Cancer. 2006 Aug 15;107(4):661-7. doi: 10.1002/cncr.22074. PMID 17024757
- [Result] Harlow SP, Krag DN, Julian TB, Ashikaga T, Weaver DL, Feldman SA, Klimberg VS, Kusminsky R, Moffat FL Jr, Noyes RD, Beitsch PD. Prerandomization Surgical Training for the National Surgical Adjuvant Breast and Bowel Project (NSABP) B-32 trial: a randomized phase III clinical trial to compare sentinel node resection to conventional axillary dissection in clinically node-negative breast cancer. Ann Surg. 2005 Jan;241(1):48-54. doi: 10.1097/01.sla.0000149429.39656.94. PMID 15621990
- [Derived] Weaver DL, Ashikaga T, Krag DN, Skelly JM, Anderson SJ, Harlow SP, Julian TB, Mamounas EP, Wolmark N. Effect of occult metastases on survival in node-negative breast cancer. N Engl J Med. 2011 Feb 3;364(5):412-21. doi: 10.1056/NEJMoa1008108. Epub 2011 Jan 19. PMID 21247310
- [Derived] Krag DN, Anderson SJ, Julian TB, Brown AM, Harlow SP, Costantino JP, Ashikaga T, Weaver DL, Mamounas EP, Jalovec LM, Frazier TG, Noyes RD, Robidoux A, Scarth HM, Wolmark N. Sentinel-lymph-node resection compared with conventional axillary-lymph-node dissection in clinically node-negative patients with breast cancer: overall survival findings from the NSABP B-32 randomised phase 3 trial. Lancet Oncol. 2010 Oct;11(10):927-33. doi: 10.1016/S1470-2045(10)70207-2. PMID 20863759

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I: Conventional Axillary Dissection | Arm II: Sentinel Node Resection Followed by Node Examination
Started | 2807 | 2804
Completed | 1975 | 2011
Not Completed | 832 | 793
Not completed — No follow up data | 3 | 0
Not completed — Sentinel node positive patients | 829 | 793

BASELINE CHARACTERISTICS:
Groups:
- Conventional Axillary Dissection: Sentinel Node Resection Followed by Conventional Axillary Dissection
- Sentinel Node Resection Followed by Node Examination: Sentinel node resection followed by node examination
- Total: Total of all reporting groups
Arm/Group | Conventional Axillary Dissection | Sentinel Node Resection Followed by Node Examination | Total
Number analyzed (Participants) | 2807 | 2804 | 5611
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (11.2) | 56 (11.0) | 56 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2807 | 2804 | 5611
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Morbidity - Number of Participants With Residual Shoulder Abduction Deficit
Description: Morbidity as measured by residual shoulder abduction deficit. Shoulder Abduction Deficit definition: Shoulder range of motion decreased by greater than or equal to 10% as compared with that measured prior to surgery.
Time Frame: Before and after surgery (within 30 days of randomization)
Population: Data missing or unknown for some patients
Measure: Count of Participants; unit: Participants
Groups:
- Arm I:Sentinel Node Resection+Conventional Axillary Dissection: Sentinel node resection immediately followed by axillary dissection
  conventional surgery: Sentinel node resection immediately followed by axillary dissection.
Arm/Group | Arm I:Sentinel Node Resection+Conventional Axillary Dissection | Arm II: Sentinel Node Resection Followed by Node Examination
Number analyzed (Participants) | 1449 | 1519
Participants | 276 | 200

2. Primary Outcome: Morbidity - Number of Participants With Residual Arm Volume Difference
Description: Morbidity as measured by residual arm volume difference. Residual Arm Volume Difference definition: Arm volume differences greater than or equal to 10% as compared with that measured prior to surgery
Time Frame: before and after surgery (within 30 days of randomization)
Population: Data missing or unknown for some patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I:Sentinel Node Resection+Conventional Axillary Dissection | Arm II: Sentinel Node Resection Followed by Node Examination
Number analyzed (Participants) | 1136 | 1151
Participants | 314 | 192

3. Primary Outcome: Morbidity - Number of Participants With Residual Arm Numbness
Description: Morbidity as measured by residual arm numbness
Time Frame: before and after surgery (within 30 days of randomization)
Population: Data missing or unknown for some patients
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I:Sentinel Node Resection+Conventional Axillary Dissection | Arm II: Sentinel Node Resection Followed by Node Examination
Number analyzed (Participants) | 1336 | 1371
Participants | 408 | 103

4. Primary Outcome: Morbidity - Number of Participants With Residual Arm Tingling
Description: Morbidity as measured by residual arm tingling
Time Frame: before and after surgery (within 30 days of randomization)
Population: Data missing or unknown for some patients
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I:Sentinel Node Resection+Conventional Axillary Dissection | Arm II: Sentinel Node Resection Followed by Node Examination
Number analyzed (Participants) | 1329 | 1343
Participants | 175 | 90

5. Primary Outcome: Overall Survival
Description: Measured at the time from randomization to any death to determine the percentage of patients alive at 8 years
Time Frame: 8 years
Population: Data missing or unknown for some patients
Measure: Number (95% Confidence Interval); unit: percentage of patients alive at 8 years
Arm/Group | Arm I:Sentinel Node Resection+Conventional Axillary Dissection | Arm II: Sentinel Node Resection Followed by Node Examination
Number analyzed (Participants) | 1975 | 2011
percentage of patients alive at 8 years | 91.8 [90.4 to 93.3] | 90.3 [88.8 to 91.8]

6. Primary Outcome: Disease-free Survival as Measured by Breast Cancer Recurrence, Any Second Primary Cancer, and Death From Any Cause in Patients Without a Prior Event.
Description: Measured at time from randomization to recurrence, second primary, or death to determine the percentage of patients disease free at 8 years.
Time Frame: 8 years
Measure: Number (95% Confidence Interval); unit: percentage pts disease free at 8 years
Arm/Group | Arm I:Sentinel Node Resection+Conventional Axillary Dissection | Arm II: Sentinel Node Resection Followed by Node Examination
Number analyzed (Participants) | 1975 | 2011
percentage pts disease free at 8 years | 82.4 [80.5 to 84.4] | 81.5 [79.6 to 83.4]

7. Secondary Outcome: Pathology Investigation of Sentinel Nodes in Sentinel Node Negative Patients to Identify a Group Who Were Potentially at Increased Risk of Systemic Recurrence
Description: Percentage of patients distant disease-free at 5 years. Sentinel node definition: Sentinel nodes are the first few lymph nodes into which a tumor drains. Sentinel node biopsy requires injecting a tracer material to help a surgeon locate sentinel nodes during surgery.
Time Frame: From the time of randomization until 5 years
Population: Data missing or unknown for some patients.
Measure: Number; unit: percentage of patients
Groups:
- Group 1: Negative Node Patients Without Occult Metastases: Patients with initially negative sentinel node tumors blocks whose tumors, upon re-examination, were not found to have had occult metastases
- Group 2: Negative Node Patients With Occult Metastases: Patients with initially negative sentinel node tumor blocks whose tumors, upon re-examination, were found to have had occult metastases
Arm/Group | Group 1: Negative Node Patients Without Occult Metastases | Group 2: Negative Node Patients With Occult Metastases
Number analyzed (Participants) | 3122 | 584
percentage of patients | 92.5 | 89.7

8. Secondary Outcome: Pathology Investigation of Sentinel Nodes in Sentinel Node Negative Patients to Identify a Group Who Were Potentially at Increased Risk of Systemic Recurrence
Description: Measured at time from randomization to any distant cancer or death to determine percentage of patients distant disease free at 5 years. Sentinel node definition: Sentinel nodes are the first few lymph nodes into which a tumor drains. Sentinel node biopsy requires injecting a tracer material to help a surgeon locate sentinel nodes during surgery.
Time Frame: From the time of randomization until 5 years
Population: Data missing or unknown for some patients
Measure: Number; unit: percentage distant disease free at 5 yrs
Arm/Group | Group 1: Negative Node Patients Without Occult Metastases | Group 2: Negative Node Patients With Occult Metastases
Number analyzed (Participants) | 3122 | 584
percentage distant disease free at 5 yrs | 92.5 | 89.7

9. Secondary Outcome: The Percentage of Technically Successful Sentinel Node Resections as Measured by the Proportion of Patients for Whom at Least One Sentinel Node is Identified.
Description: Sentinel node definition: Sentinel nodes are the first few lymph nodes into which a tumor drains. Sentinel node biopsy requires injecting a tracer material to help a surgeon locate sentinel nodes during surgery.
Time Frame: At time of surgery (within 30 days of randomization)
Population: Data missing or unknown for some patients. In Arm I, 19 patients did not accept the protocol and another 42 patients did not have a SLN resection leaving 2746 with a SLN resection. In Arm II, 4 declined the protocol treatment and another 10 patients did not have a SLN resection leaving 2790 with a SLN resection.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I:Sentinel Node Resection+Conventional Axillary Dissection | Arm II: Sentinel Node Resection Followed by Node Examination
Number analyzed (Participants) | 2746 | 2790
Participants
  Success | 2672 | 2707
  Failure | 74 | 83

10. Secondary Outcome: Sensitivity of the Sentinel Node to Determine Presence of Nodal Metastases.
Description: as for outcome 9
Time Frame: At time of surgery (within 30 days of randomization)
Population: Data not collected for some patients. This analysis as pre-specified in the approved B-32 protocol required that both a SLN resection and an ALND be performed. The patients in Arm II were assigned to have no ALND so were excluded from the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I:Sentinel Node Resection+Conventional Axillary Dissection | Arm II: Sentinel Node Resection Followed by Node Examination
Number analyzed (Participants) | 766 | 0
Participants
  False Negative | 75 |
  True Negative | 691 |

ADVERSE EVENTS:
Description: Participants at Risk includes any patient who submitted an AE form.
Groups:
- Conventional Axillary Dissection: Conventional axillary dissection
Arm/Group | Conventional Axillary Dissection | Sentinel Node Resection Followed by Node Examination
All-Cause Mortality (participants affected / at risk) | 0/2788 | 1/2800
Serious Adverse Events (participants affected / at risk) | 9/2788 | 8/2800
Other Adverse Events (participants affected / at risk) | 0/2788 | 0/2800
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Conventional Axillary Dissection (N=2788) | Sentinel Node Resection Followed by Node Examination (N=2800)
Anaphylaxis (Immune system disorders) | 5 | 5
Infections and infestations - Other, specify (Infections and infestations) | 2 | 0
Nervous system disorders - Other, specify (Nervous system disorders) | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Thromboembolic event (Vascular disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less